CLINICAL TRIAL: NCT00509119
Title: Retrospective ICP Waveform Analysis in Stroke Patients Followed Prospectively
Brief Title: ICP Waveform Analysis in Stroke Patients
Status: Withdrawn | Type: Observational
Why Stopped: Change of workplace for leading investigator, not replaced
Sponsor: Oslo University Hospital (Other)
Responsible Party: Gunnar Bentsen / Consultant, Rikshospitalet-Radiumhospitalet HF
Other Study IDs: 1-engum
Record Dates: First submitted 2007-07-30; First posted 2007-07-31 (Estimated); Last update posted 2015-04-27 (Estimated); Status verified 2010-10

CONDITIONS: Stroke
Keywords: apoplexia; Intracranial and intraarterial pressure curves in acute apoplectic patients
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a study on how acute clinical state and final clinical outcome in patients with stroke (exclusive subarachnoid hemorrhage) relate to ICP/ABP-derived pressure waveform parameters recorded during intensive care management.

DETAILED DESCRIPTION:
Aim of study:

* Prospectively collect clinical and radiological data as well as management data.
* Perform retrospective analysis of ICP/ABP recordings (mean ICP, mean ICP wave amplitude, mean ABP, mean ABP wave amplitude, CPP)
* Relate the prospectively collected data with results of retrospective pressure analysis.

ELIGIBILITY:
Inclusion Criteria:

* Acute apoplexy

Exclusion Criteria:

* Subarachnoidal bleeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute ICH
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2006-12; Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Clinical outcome | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Gunnar Bentsen, MD, Principal Investigator — Oslo University Hospital
Locations (1):
- Rikshospitalet - Radiumhospitalet HF, Oslo, Norway